CLINICAL TRIAL: NCT01857492
Title: tDCS for the Management of Chronic Visceral Pain in Patients With Chronic Pancreatitis
Acronym: tDCS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inactive
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Steven Freedman, MD PhD Professor of Medicine Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-P-000033
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Pancreatitis; Pain
Keywords: abdominal pain; pancreatitis; chronic abdominal pain; visceral pain; meditation; tDCS; noninvasive brain stimulation; EEG; Kirtan Kriya
MeSH Terms: conditions — Pancreatitis, Chronic; Pain; Abdominal Pain; Pancreatitis; Visceral Pain | interventions — Transcranial Direct Current Stimulation; Meditation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHAM (Sham Comparator): We will apply sham tDCS on the primary motor cortex. We will use the same montage and parameters of active tDCS. However the current will be applied for 30 seconds in the beginning of the procedure and after that the current is turned off. This parameter for sham stimulation was chosen based on previous studies that have shown that perceived sensations on the scalp such as tingling usually fade out in the first 30 seconds of tDCS. It should be noted that less than 3 minutes of tDCS induces no effects on cortical excitability [29] and also using 30 seconds of sham is a reliable method of blinding as shown by a randomized controlled study [30]. Subjects will also meditate while receiving stimulation
  Interventions: Device: tDCS; Behavioral: Meditation
- ACTIVE (Active Comparator): A 1x1 Low-intensity DC Stimulator such as the Soterix Medical Inc. (Model 1224-B New York, NY, USA) or an equivalent device will be used to deliver direct current through 35cm² saline-soaked electrodes. The anodal electrode will be placed over the left primary motor cortex (M1) while the cathodal electrode will be placed over the contralateral supra-orbital area. Primary motor cortex will be localized using the 10/20 EEG system (C3 or C4) and this is a reliable method for the technique of tDCS [5]. During active tDCS, a 2mA constant current will be delivered for 20 minutes while the subject meditates. The primary motor cortex is a reliable "entry port" to modulate dysfunctional activity in pain-related neural networks.
  Interventions: Device: tDCS; Behavioral: Meditation

INTERVENTIONS:
Device: tDCS
  Other Names: Soterix Medical Inc.
Behavioral: Meditation — Both Active and SHAM groups will receive Meditation.
  Other Names: Kirtan kriya Meditation

SUMMARY:
This study is testing whether the addition of a noninvasive form of brain stimulation called transcranial direct current stimulation (tDCS) when combined with meditation helps decrease the abdominal pain in patients with chronic pancreatitis. The device involved in this study, transcranial direct current stimulation (tDCS) is investigational. This means that the study device is still being tested in research studies and is not approved by the Food and Drug Administration [FDA].

DETAILED DESCRIPTION:
This is a double-blind, pilot study with the goal of testing the effects of tDCS coupled with meditation in the management of visceral pain in patients with chronic pancreatitis. We will enroll a total of 14 subjects with chronic pancreatitis. After enrollment, subjects will be randomized to active stimulation plus mediation (7 subjects) or sham stimulation plus meditation (7 subjects). Subjects will undergo 5 days of active tDCS stimulation plus meditation or sham tDCS plus meditation. Sessions will last approximately 30 min - 1 hour. EEG activity will be measured in the first, last and follow-up visits. After each stimulation session, we will assess for adverse effects using the tDCS adverse effects questionnaire. We will also have the subject fill out a pain/medication diary during the 5 days of treatment. All study procedures will be completed at BIDMC.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent to participate in the study
2. 18 years old
3. If taking pain medications, stable doses are required for at least 1 month prior to initiation of the study

Exclusion Criteria:

1. History of alcohol or substance abuse within the last 6 months as self-reported
2. Suffering from severe depression (with a score of >30 in the Beck Depression Inventory)
3. Diagnosis of any neurological diseases (such as epilepsy)
4. Episodes of seizures within the last 6 months
5. Unexplained loss of consciousness
6. Use of carbamazepine or neuropsychotropic drugs
7. Have had no neurosurgery as self reported
8. Contraindications to tDCS

   1. Metal in the head
   2. Implanted brain medical devices
9. Pregnant at time of enrollment
10. Previous experience with meditation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pain | Two weeks
  Assess the effects of 5 days of active vs sham tDCS stimulation plus meditation on chronic visceral pain in patients with chronic pancreatitis. We will determine the magnitude of pain reduction using the Visual Analog Scale (VAS) score and Brief Pain Inventory (BPI). We hypothesize that active tDCS plus meditation will have a greater decrease in VAS scores and BPI scores when compared to sham tDCS plus meditation in subjects with chronic pancreatitis

SECONDARY OUTCOMES:
Quality of Life | Two weeks
  Assess the effects of 5 days of active vs sham tDCS stimulation plus meditation on life satisfaction in subjects with chronic pancreatitis. We will use the Quality of Life Scale (QoLS) to assess changes in life satisfaction after active tDCS plus meditation intervention. We hypothesize that active tDCS plus meditation will have a greater increase in the QoLS after the intervention when compared to sham tDCS plus mediation in subjects with chronic pancreatitis

OTHER OUTCOMES:
neurophysiological measures (EEG) | Two weeks
  Determine whether treatment with active tDCS coupled with meditation changes cortical activity as assessed with electroencephalography (EEG). We hypothesize that active tDCS plus meditation will have a greater increase in alpha activity and a greater inhibition in beta activity and this will be associated with a greater reduction in pain when compared to sham tDCS plus meditation in patients with chronic pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Freedman, MD PhD, Principal Investigator — Beth Israel Deaconess Medical Center; Steven D. Freedman, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Fregni F, Potvin K, Dasilva D, Wang X, Lenkinski RE, Freedman SD, Pascual-Leone A. Clinical effects and brain metabolic correlates in non-invasive cortical neuromodulation for visceral pain. Eur J Pain. 2011 Jan;15(1):53-60. doi: 10.1016/j.ejpain.2010.08.002. Epub 2010 Sep 6. PMID 20822942
- [Background] Fregni F, DaSilva D, Potvin K, Ramos-Estebanez C, Cohen D, Pascual-Leone A, Freedman SD. Treatment of chronic visceral pain with brain stimulation. Ann Neurol. 2005 Dec;58(6):971-2. doi: 10.1002/ana.20651. No abstract available. PMID 16315281
- See also: Pancreas Center at Beth Israel Deaconess Medical Center — http://www.bidmc.org/Centers-and-Departments/Departments/Digestive-Disease-Center/Pancreas-Center.aspx